CLINICAL TRIAL: NCT01772823
Title: Project PrEPare - An Open Label Demonstration Project and Phase II Safety Study of Pre-Exposure Prophylaxis Use Among Young Men Who Have Sex With Men (YMSM) in the United States
Brief Title: An Open Label Demonstration Project and Phase II Safety Study of Pre-Exposure Prophylaxis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATN 110 Version 3.0
Record Dates: First submitted 2012-12-21; First posted 2013-01-21 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-12

CONDITIONS: HIV Infection
Keywords: HIV, PrEP, FTC/TDF, Truvada®
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 3MV Behavioral Intervention Group (Experimental): 3MV Behavioral Intervention combined with open label FTC/TDF (Truvada®) as PrEP
  Interventions: Behavioral: 3MV; Drug: Emtricitabine/tenofovir (FTC/TDF (Truvada®))
- PCC Behavioral Intervention Group (Experimental): PCC Behavioral Intervention combined with open label FTC/TDF (Truvada®) as PrEP
  Interventions: Behavioral: PCC; Drug: Emtricitabine/tenofovir (FTC/TDF (Truvada®))

INTERVENTIONS:
Behavioral: 3MV — Many Men, Many Voices (3MV) is based on Social Cognitive Theory and the Transtheoretical Model of Behavior Change. 3MV is a group-level intervention that addresses behavioral and social determinants and other factors influencing the HIV/sexually transmitted infection (STI) risk and protective behaviors of Men having sex with men (MSM) of color. The other factors include cultural, social and religious norms, racial identity and degree of connectedness to communities, HIV/STI interactions, sexual relationship dynamics, and the social influences of racism and homophobia.
  Other Names: Many Men, Many Voices
  Arms: 3MV Behavioral Intervention Group
Behavioral: PCC — Personalized Cognitive Counseling (PCC) is based on the Model of Relapse Prevention and Gold's Self-Appraisal of Risk Behavior. PCC is a 1-hour, single-session, individual level intervention administered by a trained counselor in a clinic setting. Counselors ask the client to recall and describe in as much detail, a recent encounter of unprotected anal sex with another man of unknown or sero-discordant HIV status. The client then identifies and expresses thoughts, feelings, or attitudes that might have led to the high-risk behavior. The client and counselor examine and identify thoughts that may have led the client to decide to engage in high transmission risk sex. The client and counselor agree on strategies that can be used to deal with similar situations in the future.
  Other Names: Personalized Cognitive Counseling
  Arms: PCC Behavioral Intervention Group
Drug: Emtricitabine/tenofovir (FTC/TDF (Truvada®)) — All subjects will be provided with daily FTC/TDF (Truvada®) as Pre-exposure prophylaxis (PrEP) for 48 weeks.
  Other Names: FTC/TDF; Truvada®; Emtricitabine/tenofovir; PrEP

SUMMARY:
Approximately 200 HIV-uninfected young men who have sex with men (YMSM) at high risk of acquiring HIV infection, ages 18-22 years, inclusive, will be recruited across all participating Adolescent Medicine Trials Units (AMTU). The behavioral intervention will be assigned at the level of the site, which include Many Men, Many Voices (3MV) and Personalized Cognitive Counseling (PCC). Subjects will first complete the behavioral intervention offered at their respective site and then be provided with open label emtricitabine (FTC)/tenofovir (TDF) (Truvada®) as PrEP. Behavioral and biomedical data will be collected at baseline and 0, 4, 8, 12, 24, 36 and 48 weeks. Any subjects who become HIV infected during the course of the study will be discontinued from the study agent and followed for an additional 24 weeks after the study visit at which HIV infection is confirmed. Those subjects who meet specific bone or renal criteria at the Week 48 visit or the 24-Week HIV Seropositive visit will be followed for an additional 48 weeks in the Extension Phase to monitor longer-term outcomes of potential concerns.

DETAILED DESCRIPTION:
The primary objectives of the study are to provide additional safety data regarding FTC/TDF (Truvada®) use as PrEP in YMSM, to examine acceptability, patterns of use, rates of adherence, measure levels of drug exposure and patterns of risk behavior when YMSM are provided open label FTC/TDF (Truvada®). The study will also examine information regarding safety and efficacy of FTC/TDF (Truvada®) as PrEP from prior studies.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent;
* Male gender at birth;
* Age 18 years and 0 days through 22 years and 364 days, inclusive, at the time of signed informed consent;
* Self reports evidence of high risk for acquiring HIV infection including at least one of the following:

  * At least one episode of unprotected anal intercourse with an HIV-infected male partner or a male partner of unknown HIV status during the last 6 months;
  * Anal intercourse with 3 or more male sex partners during the last 6 months;
  * Exchange of money, gifts, shelter, or drugs for anal sex with a male partner during the last 6 months;
  * Sex with a male partner and has had a sexually transmitted infection (STI) during the last 6 months or at screening;
  * Sexual partner of an HIV-infected man with whom condoms were not consistently used in the last 6 months; or
  * At least one episode of anal intercourse where the condom broke or slipped off during the last 6 months;
* Tests HIV antibody negative at time of screening;
* Willing to provide locator information to study staff;
* Willing to take pre-exposure prophylaxis (PrEP);
* Willing to participate in behavioral intervention;
* Reports intention not to relocate out of the Adolescent Medicine Trial Unit (AMTU) study area during the course of the study; and
* Does not have a job or other obligations that would require long absences from the AMTU study area (greater than 4 weeks at a time).

Exclusion Criteria:

* Appears visibly distraught or presence of active serious psychiatric symptoms (e.g., active hallucinations, suicidal, homicidal, or exhibiting violent behavior) at the time of consent;
* Intoxicated or under the influence of alcohol or other drugs at the time of consent;
* Any significant uncontrolled, active or chronic disease process that, in the judgment of the site investigator, would make participation in the study inappropriate. (Appropriately managed conditions, like well-controlled diabetes, would not preclude enrollment; the site is encouraged to contact the Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) 110 Protocol Team if they are having difficulty making the judgment.);
* History of bone fractures not explained by trauma;
* Acute or chronic hepatitis B infection as indicated by positive hepatitis B surface antigen (sAg) test at time of screening;
* Confirmed renal dysfunction (Creatinine Clearance (CrCl) < 75 ml/min, or serum creatinine ≥ upper limit of normal (ULN), or history of renal parenchymal disease or presence of only one kidney at time of screening;
* Confirmed ≥ Grade 2 hypophosphatemia at time of screening;
* Confirmed ≥ Grade 2 hematologic system abnormality (White Blood Count (WBC), Absolute Neutrophil Count (ANC), hemoglobin, or platelets) at time of screening;
* Confirmed ≥ Grade 2 hepatobiliary system abnormality (Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), or bilirubin) at time of screening;
* Confirmed proteinuria as indicated by urine dipstick result ≥ 1+ at time of screening, regardless of urine protein to creatinine ratio(UP/C);
* UP/C > 0.37 g/g at time of screening, regardless of urine dipstick protein result;
* Confirmed normoglycemic glucosuria as indicated by urine dipstick result ≥ 1+ in the presence of normal serum glucose (<120 mg/dL) at time of screening;
* A confirmed Grade ≥ 3 toxicity on any screening evaluations;
* Known allergy/sensitivity to the study agent or its components;
* Concurrent participation in an HIV vaccine study or other investigational drug study, including oral or topical PrEP (microbicide) studies;
* Use of disallowed medications ; or
* Inability to understand spoken English.

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sybil Hosek, PhD, Study Chair — Cook County Health & Hospitals System
Locations (12):
- United States (12):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Colorado - The Children's Hospital of Denver, Aurora, Colorado
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stroger Hospital and the CORE Center, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Fenway Institute, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Childrens Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Havens PL, Perumean-Chaney SE, Patki A, Cofield SS, Wilson CM, Liu N, Anderson PL, Landovitz RJ, Kapogiannis BG, Hosek SG, Mulligan K. Changes in Bone Mass After Discontinuation of Preexposure Prophylaxis With Tenofovir Disoproxil Fumarate/Emtricitabine in Young Men Who Have Sex With Men: Extension Phase Results of Adolescent Trials Network Protocols 110 and 113. Clin Infect Dis. 2020 Feb 3;70(4):687-691. doi: 10.1093/cid/ciz486. PMID 31179503
- [Derived] Castillo-Mancilla J, Seifert S, Campbell K, Coleman S, McAllister K, Zheng JH, Gardner EM, Liu A, Glidden DV, Grant R, Hosek S, Wilson CM, Bushman LR, MaWhinney S, Anderson PL. Emtricitabine-Triphosphate in Dried Blood Spots as a Marker of Recent Dosing. Antimicrob Agents Chemother. 2016 Oct 21;60(11):6692-6697. doi: 10.1128/AAC.01017-16. Print 2016 Nov. PMID 27572401
- See also: ATN website — http://www.atnonline.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This research was conducted at 12 clinical sites. Accrual was open between July 2012 and September 2013.
Groups:
- 3MV Behavioral Intervention Group: 3MV is a group-level intervention that addresses behavioral and social determinants and other factors influencing the HIV/sexually transmitted infection (STI) risk and protective behaviors of Men having sex with men (MSM) of color. The 3MV intervention was conducted as a 2-day seminar with approximately 10-20 subjects per sessions. After completion of the 3MV intervention, all subjects were provided with daily FTC/TDF (Truvada®) as Pre-exposure prophylaxis (PrEP) for 48 weeks.
- PCC Behavioral Intervention Group: PCC is based on the Model of Relapse Prevention and Gold's Self-Appraisal of Risk Behavior. The PCC intervention was conducted as a 1-hour, single-session, individual level intervention administered by a trained counselor in a clinic setting. After completion of the PCC intervention, all subjects were provided with daily FTC/TDF (Truvada®) as Pre-exposure prophylaxis (PrEP) for 48 weeks.
Period: Behavioral Intervention (BL -3MV or PCC)
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Started | 128 | 72
Completed | 116 | 70
Not Completed | 12 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Inadvertent enrollment | 1 | 0
Not completed — Inelligible at rescreen | 2 | 1
Not completed — Wk 0 not completed, 30 days of baseline | 6 | 0
Not completed — Moved out of area | 1 | 0
Period: Treatment Phase (Week 0- Week 48)
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Started | 116 | 70
Completed | 88 | 52
Not Completed | 28 | 18
Not completed — Lost to Follow-up | 15 | 13
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Moved out of area | 4 | 3
Not completed — Incarcerated | 1 | 0
Not completed — Suicide gesture/disruptive behavior | 1 | 0
Not completed — Wk 0 not completed, 30 days of baseline | 1 | 1
Period: Extension Phase (Visits 24,48wks Post tx
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Started | 63 (25 of the 88 subjects that completed the Treatment Phase were not eligible for the Extension Phase) | 42 (10 of the 52 subjects that completed the Treatment Phase were not eligible for the Extension Phase)
Completed | 53 | 33
Not Completed | 10 | 9
Not completed — Lost to Follow-up | 6 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Moved out of area | 2 | 2
Not completed — Became unavailable for study visits | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group | Total
Number analyzed (Participants) | 128 | 72 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.14 (1.40) | 20.25 (1.23) | 20.18 (1.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 128 | 72 | 200
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Asian/Pacific Islander | 2 | 0 | 2
  Race/ethnicity: Black/African American | 55 | 38 | 93
  Race/ethnicity: White | 26 | 16 | 42
  Race/ethnicity: White/Hispanic | 15 | 6 | 21
  Race/ethnicity: Other/Mixed Race | 30 | 12 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic Ethnicity: Hispanic | 39 | 14 | 53
  Hispanic Ethnicity: Non-Hispanic | 89 | 56 | 145
  Hispanic Ethnicity: Refused | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 128 | 72 | 200
BMI [Count of Participants; unit: Participants]
  Underweight (<18.5 kg/m^2) | 3 | 6 | 9
  Normal (18.5-<25 kg/m^2) | 71 | 38 | 109
  Overweight (25.0-<30 kg/m^2) | 25 | 18 | 43
  Obese (=>30 kg/m^2) | 29 | 10 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serum Creatinine Event of Grade 1 or Higher
Description: This measure addresses the objective: Additional safety data regarding FTC/TDF (Truvada®) use among HIV-uninfected YMSM
  Serum creatinine was tested at every study visit (Baseline through Week 48). The number of participants with a serum creatinine laboratory toxicity of Grade 1 or higher was assessed. Grade 1 (Mild) toxicity was defined as: 1.1 - 1.3 x ULN, where ULN is the Upper limit of normal.
Time Frame: 48 Weeks
Population: Participants with visit data through 48 weeks. The primary objective "Additional safety data regarding FTC/TDF (Truvada®) use" did not involve comparison of the behavioral intervention groups. All participants in both groups received FTC/TDF (Truvada®). As a result, this outcome was not assessed separately for each group.
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants: Combined data for all participants that participated in either the 3MV or PCC arms/groups as part of the study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 137
Participants | 1

2. Primary Outcome: Number of Participants With Decrease in Absolute Bone Mineral Density (BMD) From Baseline to Week 48
Description: This outcome addresses the objective "Additional Safety Data Regarding FTC/TDF (Truvada®) Use Among HIV-uninfected YMSM."
  The total number of participants with dual-energy radiography absorptiometry scanning (DXA) data through Week 48 who experienced varying degrees of decrease in absolute BMD in at least one region (spine, hip, or whole body) between Baseline and Week 48.
Time Frame: 48 weeks
Population: Enrolled subjects with DXA results for Baseline and Week 48 The primary objective "Additional safety data regarding FTC/TDF (Truvada®) use" did not involve comparison of the behavioral intervention groups. All participants in both groups received FTC/TDF (Truvada®). As a result, this outcome was not assessed separately for each group.
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 135
Participants
  Decrease in absolute BMD >=1% | 97
  Decrease in absolute BMD >=5% | 16
  Decrease in absolute BMD >10% | 1

3. Primary Outcome: Lumbar Spine Bone Mineral Density at Baseline and at Week 48
Description: This outcome addresses the objective: Additional Safety Data Regarding FTC/TDF (Truvada®) Use Among HIV-uninfected YMSM.
  Bone mineral density at Baseline and Week 48: data reported below for lumbar spine.
Time Frame: Baseline, Week 48
Population: Participants with DXA results. (Baseline N=197, Week 48 N=135). The primary objective "Additional safety data regarding FTC/TDF (Truvada®) use" does not involve comparison of the behavioral intervention groups. All participants in both groups received FTC/TDF (Truvada®). As a result, this outcome was not assessed separately for each group.
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | All Study Participants
Number analyzed (Participants) | 197
g/cm2
  Lumbar spine BMD at baseline | 1.09 (0.15)
  Lumbar spine BMD Week 48: number analyzed (Participants) | 135
  Lumbar spine BMD Week 48 | 1.08 (0.14)

4. Primary Outcome: Femoral Neck Bone Mineral Density at Baseline and at Week 48
Description: This outcome addresses the objective: Additional Safety Data Regarding FTC/TDF (Truvada®) Use Among HIV-uninfected YMSM.
  Bone mineral density at Baseline and Week 48: data reported below for femoral neck.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | All Study Participants
Number analyzed (Participants) | 197
g/cm2
  Femoral neck BMD at baseline | 1.04 (0.18)
  Femoral neck Week 48: number analyzed (Participants) | 135
  Femoral neck Week 48 | 1.03 (0.20)

5. Primary Outcome: Total Body Bone Mineral Density at Baseline and at Week 48
Description: This outcome addresses the objective: Additional Safety Data Regarding FTC/TDF (Truvada®) Use Among HIV-uninfected YMSM.
  Bone mineral density at Baseline and Week 48: data reported below for total body.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | All Study Participants
Number analyzed (Participants) | 197
g/cm2
  Total body BMD at baseline | 1.20 (.011)
  Total body BMD Week 48: number analyzed (Participants) | 135
  Total body BMD Week 48 | 1.18 (0.11)

6. Primary Outcome: Total Hip Bone Mineral Density at Baseline and at Week 48
Description: This outcome addresses the objective: Additional Safety Data Regarding FTC/TDF (Truvada®) Use Among HIV-uninfected YMSM.
  Bone mineral density at Baseline and Week 48: data reported below for total hip.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | All Study Participants
Number analyzed (Participants) | 197
g/cm2
  Total hip BMD at baseline | 1.10 (0.16)
  Total hip BMD Week 48: number analyzed (Participants) | 135
  Total hip BMD Week 48 | 1.08 (0.17)

7. Primary Outcome: Number of Participants With Unprotected Sex Acts
Description: This outcome addresses the objective "Additional Safety Data Regarding FTC/TDF (Truvada®) Use Among HIV-uninfected YMSM," specifically behavioral disinhibition/risk compensation endpoints.
  Responses to the participant ACASI question referring to male partners in the past month/since the last survey:
  "Of these males (male partners), how many did you have unprotected oral or anal sex with in the last month?" (Baseline), or "Of these males (male partners), how many did you have unprotected oral or anal sex with since the last time you took this survey?" (Week 48) An event is defined as an answer of greater than 0.
Time Frame: Baseline and 48 weeks
Population: Participants at Baseline/Week 48 providing a response to this question. The primary objective "Additional safety data regarding FTC/TDF (Truvada®) use" did not involve comparison of the behavioral intervention groups. All participants in both groups received FTC/TDF (Truvada®). As a result, this outcome was not assessed separately for each group.
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 200
Participants
  Had unprotected oral/anal w/male (BL): number analyzed (Participants) | 177
  Had unprotected oral/anal w/male (BL) | 143
  Had unprotected oral/anal w/ male (Wk48): number analyzed (Participants) | 119
  Had unprotected oral/anal w/ male (Wk48) | 103

8. Primary Outcome: Number of Sex Partners
Description: This outcome addresses the objective "Additional Safety Data Regarding FTC/TDF (Truvada®) Use Among HIV-uninfected YMSM," specifically behavioral disinhibition/risk compensation endpoints.
  Responses to the participant ACASI question referring to number of male partners in the past month/since the last survey:
  "During the past month, how many male partners have you had sexual contact with (oral or anal)?" (Baseline), or "Since the last time you took this survey, how many male partners have you had sexual contact with (oral or anal)?" (Week 48)
  And responses to the participant ACASI question referring to number of HIV-positive male partners in the past month/since the last survey:
  "Of those you had unprotected sex with, how many did you know were HIV positive?"
Time Frame: Baseline and 48 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: sexual partners
Arm/Group | All Study Participants
Number analyzed (Participants) | 200
sexual partners
  Male sexual partners last month (baseline) | 5.41 (26.03)
  Male sexual partners since last survey (Wk 48): number analyzed (Participants) | 137
  Male sexual partners since last survey (Wk 48) | 2.46 (2.92)
  Number HIV+ male partners last month (baseline) | 1.65 (16.77)
  Number HIV+ male partners since last survey(Wk48): number analyzed (Participants) | 137
  Number HIV+ male partners since last survey(Wk48) | 0.15 (0.38)

9. Primary Outcome: Acceptability of PrEP: Distribution of Participant Feelings About Size of the Pill
Description: This outcome addresses the objective: Acceptability When YMSM Are Provided Open Label FTC/TDF (Truvada®) and Information Regarding the Safety and Efficacy of PrEP From Prior Studies.
  Acceptability of PrEP as measured by the acceptability assessment that includes questions on usability of PrEP, user-friendliness of the medication regimen, including an assessment of side effects and delivery format, and acceptability of behavioral intervention sessions. This question reports on how the participants felt about the size of the pill.
Time Frame: Week 12
Population: Participants enrolled at Week 12 who provided a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 101 | 61
Participants
  Did not like it at all | 13 | 5
  Did not like | 26 | 18
  Liked | 60 | 36
  Liked a lot | 2 | 2
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.7513, Chi-squared — The chi-squared test of homogeneity is used to assess whether the proportions of the independent variable (participant feelings on the "Size of the Pill") differ between intervention arms

10. Primary Outcome: Acceptability of PrEP: Distribution of Participant Feelings About Taste of the Pill
Description: This outcome addresses the objective: "Acceptability when YMSM are provided open label FTC/TDF (Truvada®) and information regarding the safety and efficacy of PrEP from prior studies"
  Acceptability of PrEP as measured by the acceptability assessment that includes questions on usability of PrEP, user-friendliness of the medication regimen, including an assessment of side effects and delivery format, and acceptability of behavioral intervention sessions.
  This specific outcome focuses on the question of how participants felt about the taste of the pill.
Time Frame: Week 12
Population: Participants enrolled at Week 12 who provided a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 100 | 61
Participants
  Did not like it at all | 11 | 8
  Did not like | 33 | 23
  Liked | 53 | 29
  Liked a lot | 3 | 1
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.8281, Chi-squared — The chi-squared test of homogeneity is used to assess whether the proportions of the independent variable (participant feelings on the "Taste of the Pill") differ between intervention arms; Pearson Chi-Square

11. Primary Outcome: Acceptability of PrEP: Distribution of Participant Feelings About Color of the Pill
Description: This outcome addresses the objective: "Acceptability when YMSM are provided open label FTC/TDF (Truvada®) and information regarding the safety and efficacy of PrEP from prior studies"
  Acceptability of PrEP as measured by the acceptability assessment that includes questions on usability of PrEP, user-friendliness of the medication regimen, including an assessment of side effects and delivery format, and acceptability of behavioral intervention sessions.
  This specific outcome focuses on the question of how participants felt about the color of the pill.
Time Frame: Week 12
Population: Participants enrolled at Week 12 who provided a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 101 | 61
Participants
  Did not like it at all | 3 | 2
  Did not like | 7 | 6
  Liked | 73 | 48
  Liked a lot | 18 | 5
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.3761, Chi-squared — The chi-squared test of homogeneity is used to assess whether the proportions of the independent variable (participant feelings on the "Color of the Pill") differ between intervention arms

12. Primary Outcome: Acceptability of PrEP: Distribution of Participant Feelings About Taking the Pill Every Day
Description: This outcome addresses the objective: "Acceptability when YMSM are provided open label FTC/TDF (Truvada®) and information regarding the safety and efficacy of PrEP from prior studies."
  Acceptability of PrEP as measured by the acceptability assessment that includes questions on usability of PrEP, user-friendliness of the medication regimen, including an assessment of side effects and delivery format, and acceptability of behavioral intervention sessions.
  This specific outcome focuses on the question of how participants felt about taking the pill every day.
Time Frame: Week 12
Population: Participants enrolled at Week 12 who provided a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 100 | 60
Participants
  Did not like it at all | 6 | 4
  Did not like | 24 | 17
  Liked | 63 | 31
  Liked a lot | 7 | 8
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.4359, Chi-squared — The chi-squared test of homogeneity is used to assess whether the proportions of the independent variable (participant feelings on "Taking the pill every day") differ between intervention arms

13. Primary Outcome: Acceptability of PrEP: Distribution of Participant Feelings About Taking Part in the Study
Description: This outcome addresses the objective "Acceptability when YMSM are provided open label FTC/TDF (Truvada®) and information regarding the safety and efficacy of PrEP from prior studies."
  Acceptability of PrEP as measured by the acceptability assessment that includes questions on usability of PrEP, user-friendliness of the medication regimen, including an assessment of side effects and delivery format, and acceptability of behavioral intervention sessions.
  This specific outcome focuses on the question of how participants felt about taking part in the study.
Time Frame: Week 12
Population: Participants enrolled at Week 12 who provided a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 102 | 61
Participants
  Did not like it at all | 1 | 1
  Did not like | 2 | 1
  Liked | 35 | 29
  Liked a lot | 64 | 30
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.3801, Chi-squared — The chi-squared test of homogeneity is used to assess whether the proportions of the independent variable (participant feelings on "Taking part in the study") differ between intervention arms

14. Primary Outcome: Acceptability of PrEP: Distribution of Participant Feelings About HIV Test at Every Visit
Description: This outcome addresses the objective: Acceptability When YMSM Are Provided Open Label FTC/TDF (Truvada®) and Information Regarding the Safety and Efficacy of PrEP From Prior Studies.
  Acceptability of PrEP as measured by the acceptability assessment that includes questions on usability of PrEP, user-friendliness of the medication regimen, including an assessment of side effects and delivery format, and acceptability of behavioral intervention sessions. This question reports on how the participants felt about having an HIV test at every visit.
Time Frame: Week 12
Population: Participants enrolled at Week 12 who provided a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 102 | 61
Participants
  Did not like it at all | 1 | 0
  Did not like | 1 | 4
  Liked | 29 | 15
  Liked a lot | 71 | 42
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.1968, Chi-squared — The chi-squared test of homogeneity is used to assess whether the proportions of the independent variable (participant feelings on "HIV test at every visit") differ between intervention arms

15. Primary Outcome: Acceptability of PrEP: Distribution of Participant Feelings About Risk Reduction Counseling at Every Visit
Description: This outcome addresses the objective: Acceptability When YMSM Are Provided Open Label FTC/TDF (Truvada®) and Information Regarding the Safety and Efficacy of PrEP From Prior Studies.
  Acceptability of PrEP as measured by the acceptability assessment that includes questions on usability of PrEP, user-friendliness of the medication regimen, including an assessment of side effects and delivery format, and acceptability of behavioral intervention sessions. This question reports on how the participants felt about having individual risk reduction counseling at every visit
Time Frame: Week 12
Population: Participants enrolled at Week 12 who provided a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 102 | 61
Participants
  Did not like it at all | 2 | 1
  Did not like | 1 | 5
  Liked | 38 | 23
  Liked a lot | 61 | 32
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.1226, Chi-squared — The chi-squared test of homogeneity is used to assess whether the proportions of the independent variable (participant feelings on "Risk Reduction counseling at every visit") differ between intervention arms

16. Primary Outcome: Acceptability of PrEP: Distribution of Participant Feelings About Questions About Sexual Behavior
Description: This outcome addresses the objective: Acceptability When YMSM Are Provided Open Label FTC/TDF (Truvada®) and Information Regarding the Safety and Efficacy of PrEP From Prior Studies.
  Acceptability of PrEP as measured by the acceptability assessment that includes questions on usability of PrEP, user-friendliness of the medication regimen, including an assessment of side effects and delivery format, and acceptability of behavioral intervention sessions. This question reports on how the participants felt about being asked questions about sexual behavior at every visit
Time Frame: Week 12
Population: Participants enrolled at Week 12 who provided a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 101 | 61
Participants
  Did not like it at all | 1 | 1
  Did not like | 8 | 13
  Liked | 61 | 31
  Liked a lot | 31 | 16
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.0994, Chi-squared — The chi-squared test of homogeneity is used to assess whether the proportions of the independent variable (participant feelings on "Questions about sexual behavior") differ between intervention arms

17. Primary Outcome: Acceptability of PrEP: Distribution of Participant Feelings About Physician Exam
Description: This outcome addresses the objective: Acceptability When YMSM Are Provided Open Label FTC/TDF (Truvada®) and Information Regarding the Safety and Efficacy of PrEP From Prior Studies.
  Acceptability of PrEP as measured by the acceptability assessment that includes questions on usability of PrEP, user-friendliness of the medication regimen, including an assessment of side effects and delivery format, and acceptability of behavioral intervention sessions. This question reports on how the participants felt about having a physician exam by a doctor
Time Frame: Week 12
Population: Participants enrolled at Week 12 who provided a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 101 | 61
Participants
  Did not like it at all | 1 | 1
  Did not like | 13 | 4
  Liked | 54 | 38
  Liked a lot | 33 | 18
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.5285, Chi-squared — The chi-squared test of homogeneity is used to assess whether the proportions of the independent variable (participant feelings on the "Physician exam") differ between intervention arms

18. Primary Outcome: Patterns of Use, Rates of Adherence and Measured Levels of Open Label FTC/TDF (Truvada®) Drug Exposure
Description: This outcome addresses the objective: "Patterns of Use, Rates of Adherence and Measured Levels of Drug Exposure When YMSM Are Provided Open Label FTC/TDF (Truvada®) and Information Regarding the Safety and Efficacy of PrEP From Prior Studies."
  PrEP medication levels were assessed via dried blood spot (DBS) collected at each visit to quantify intracellular TFV-DP and FTC-triphosphate concentrations. DBS results were translated into dosing categories previously used in PrEP trials with adult MSM. Dosing categories included below lower limit of quantitation (BLQ), lower limit of quantitation to 349 fmol per punch (fewer than 2 tablets per week), 350- 699 fmol per punch (2-3 tablets per week), 700-1250 fmol per punch (4 tablets per week), and >1250 fmol per punch (daily).
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48
Population: Enrolled subjects (Individual row Ns vary due to the number of subjects per week enrolled at that time point and with DBS data) This primary objective did not involve comparison of the behavioral intervention groups. All participants in both groups received FTC/TDF (Truvada®). As a result, this outcome was not assessed separately for each group.
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 200
Participants
  Week 4: number analyzed (Participants) | 173
  Week 4: Below level of quantification | 13
  Week 4: <2 days | 35
  Week 4: 2 days | 58
  Week 4: 4 days | 59
  Week 4: Daily | 8
  Week 8: number analyzed (Participants) | 164
  Week 8: Below level of quantification | 7
  Week 8: <2 days | 32
  Week 8: 2 days | 30
  Week 8: 4 days | 69
  Week 8: Daily | 26
  Week 12: number analyzed (Participants) | 159
  Week 12: Below level of quantification | 12
  Week 12: <2 days | 32
  Week 12: 2 days | 26
  Week 12: 4 days | 55
  Week 12: Daily | 34
  Week 24: number analyzed (Participants) | 148
  Week 24: Below level of quantification | 28
  Week 24: <2 days | 36
  Week 24: 2 days | 14
  Week 24: 4 days | 42
  Week 24: Daily | 28
  Week 36: number analyzed (Participants) | 134
  Week 36: Below level of quantification | 30
  Week 36: <2 days | 27
  Week 36: 2 days | 23
  Week 36: 4 days | 26
  Week 36: Daily | 28
  Week 48: number analyzed (Participants) | 120
  Week 48: Below level of quantification | 37
  Week 48: <2 days | 24
  Week 48: 2 days | 18
  Week 48: 4 days | 26
  Week 48: Daily | 15

19. Primary Outcome: Measured Levels of Drug Exposure (DBS RBC FTC-TP) When YMSM Are Provided Open Label FTC/TDF (Truvada®)
Description: PrEP medication levels were assessed via dried blood spot (DBS) collected at each visit to quantify intracellular FTC-triphosphate concentrations.
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: pmol/punch
Arm/Group | All Study Participants
Number analyzed (Participants) | 200
pmol/punch
  DBS RBC FTC-TP at Week 4: number analyzed (Participants) | 173
  DBS RBC FTC-TP at Week 4 | 0.20 (0.11)
  DBS RBC FTC-TP at Week 8: number analyzed (Participants) | 164
  DBS RBC FTC-TP at Week 8 | 0.19 (0.12)
  DBS RBC FTC-TP at Week 12: number analyzed (Participants) | 159
  DBS RBC FTC-TP at Week 12 | 0.18 (0.12)
  DBS RBC FTC-TP at Week 24: number analyzed (Participants) | 148
  DBS RBC FTC-TP at Week 24 | 0.16 (0.12)
  DBS RBC FTC-TP at Week 36: number analyzed (Participants) | 134
  DBS RBC FTC-TP at Week 36 | 0.17 (0.13)
  DBS RBC FTC-TP at Week 48: number analyzed (Participants) | 120
  DBS RBC FTC-TP at Week 48 | 0.15 (0.13)

20. Primary Outcome: Measured Levels of Drug Exposure (DBS RBC TFV-DP) When YMSM Are Provided Open Label FTC/TDF (Truvada®)
Description: This outcome addresses the objective: "Measured Levels of Drug Exposure (DBS RBC TFV-DP) When YMSM Are Provided Open Label FTC/TDF (Truvada®) and Information Regarding the Safety and Efficacy of PrEP From Prior Studies."
  PrEP medication levels were assessed via dried blood spot (DBS) collected at each visit to quantify intracellular TFV-DP concentrations.
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: fmol/punch
Arm/Group | All Study Participants
Number analyzed (Participants) | 200
fmol/punch
  DBS RBC TFV-DP at Week 4: number analyzed (Participants) | 173
  DBS RBC TFV-DP at Week 4 | 584.56 (365.37)
  DBS RBC TFV-DP at Week 8: number analyzed (Participants) | 164
  DBS RBC TFV-DP at Week 8 | 783.18 (505.67)
  DBS RBC TFV-DP at Week 12: number analyzed (Participants) | 159
  DBS RBC TFV-DP at Week 12 | 793.37 (548.87)
  DBS RBC TFV-DP at Week 24: number analyzed (Participants) | 148
  DBS RBC TFV-DP at Week 24 | 657.66 (619.06)
  DBS RBC TFV-DP at Week 36: number analyzed (Participants) | 134
  DBS RBC TFV-DP at Week 36 | 671.72 (678.37)
  DBS RBC TFV-DP at Week 48: number analyzed (Participants) | 120
  DBS RBC TFV-DP at Week 48 | 528.24 (570.80)

21. Secondary Outcome: Acceptability and Feasibility of Two Types of Efficacious Sexual Risk Reduction Interventions as Measured by Session Evaluation. Item 1 of 10: "I Learned a Lot From This Workshop/Session."
Description: Study subjects were given a brief Session Evaluation Form at the end of the behavioral intervention session consisting of ten items on a 4-point response scale aimed at eliciting information about the subject's experience with the session (i.e., was the session interesting, was it relevant to their life, did they learn from the session).
  Item 1 of 10: "I learned a lot from this workshop/session"
Time Frame: 48 weeks
Population: Participants providing a response to this question on the Session Evaluation Form
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 68 | 83
Participants
  Strongly agree | 47 | 32
  Agree | 16 | 47
  Disagree | 2 | 4
  Strongly Disagree | 3 | 0
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.0001, Chi-squared — The chi-squared test of homogeneity is used to assess whether the proportions of the independent variable (participant responses to the session evaluation question) differ between intervention arms

22. Secondary Outcome: Acceptability and Feasibility of Two Types of Efficacious Sexual Risk Reduction Interventions as Measured by Session Evaluation. Item 2 of 10: "I Will be Able to Apply What I Learned From This Workshop/Session in my Life."
Description: Study subjects were given a brief Session Evaluation Form at the end of the behavioral intervention session consisting of ten items on a 4-point response scale aimed at eliciting information about the subject's experience with the session (i.e., was the session interesting, was it relevant to their life, did they learn from the session).
  Item 2 of 10: "I will be able to apply what I learned from this workshop/session in my life"
Time Frame: 48 weeks
Population: Participants providing a response to this question on the Session Evaluation Form
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 68 | 83
Participants
  Strongly agree | 50 | 48
  Agree | 13 | 34
  Disagree | 2 | 1
  Strongly Disagree | 3 | 0
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.0098, Chi-squared — [p-value comment as in outcome 21, analysis 1]

23. Secondary Outcome: Acceptability and Feasibility of Two Types of Efficacious Sexual Risk Reduction Interventions as Measured by Session Evaluation. Item 3 of 10: "I Was Given an Opportunity to Participate and Discuss Information With Others."
Description: Study subjects were given a brief Session Evaluation Form at the end of the behavioral intervention session consisting of ten items on a 4-point response scale aimed at eliciting information about the subject's experience with the session (i.e., was the session interesting, was it relevant to their life, did they learn from the session).
  Item 3 of 10: "I was given an opportunity to participate and discuss information with others"
Time Frame: 48 weeks
Population: Participants providing a response to this question on the Session Evaluation Form
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 68 | 82
Participants
  Strongly agree | 55 | 55
  Agree | 10 | 21
  Disagree | 0 | 4
  Strongly Disagree | 3 | 2
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.0766, Chi-squared — [p-value comment as in outcome 21, analysis 1]

24. Secondary Outcome: Acceptability and Feasibility of Two Types of Efficacious Sexual Risk Reduction Interventions as Measured by Session Evaluation. Item 4 of 10: "The Workshop/Session Was Well Organized."
Description: Study subjects were given a brief Session Evaluation Form at the end of the behavioral intervention session consisting of ten items on a 4-point response scale aimed at eliciting information about the subject's experience with the session (i.e., was the session interesting, was it relevant to their life, did they learn from the session).
  Item 4 of 10: "The workshop/session was well organized"
Time Frame: 48 weeks
Population: Participants providing a response to this question on the Session Evaluation Form
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 68 | 82
Participants
  Strongly agree | 49 | 66
  Agree | 13 | 15
  Disagree | 4 | 1
  Strongly Disagree | 2 | 0
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.1581, Chi-squared — [p-value comment as in outcome 21, analysis 1]

25. Secondary Outcome: Acceptability and Feasibility of Two Types of Efficacious Sexual Risk Reduction Interventions as Measured by Session Evaluation. Item 5 of 10: "The Topic of This Workshop/Session Was Interesting."
Description: Study subjects were given a brief Session Evaluation Form at the end of the behavioral intervention session consisting of ten items on a 4-point response scale aimed at eliciting information about the subject's experience with the session (i.e., was the session interesting, was it relevant to their life, did they learn from the session).
  Item 5 of 10: "The topic of this workshop/session was interesting"
Time Frame: 48 weeks
Population: Participants providing a response to this question on the Session Evaluation Form
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 67 | 82
Participants
  Strongly agree | 47 | 56
  Agree | 16 | 23
  Disagree | 2 | 3
  Strongly Disagree | 2 | 0
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.4300, Chi-squared — [p-value comment as in outcome 21, analysis 1]

26. Secondary Outcome: Acceptability and Feasibility of Two Types of Efficacious Sexual Risk Reduction Interventions as Measured by Session Evaluation. Item 6 of 10: "The Presenter(s) Stimulated my Interest in the Material."
Description: Study subjects were given a brief Session Evaluation Form at the end of the behavioral intervention session consisting of ten items on a 4-point response scale aimed at eliciting information about the subject's experience with the session (i.e., was the session interesting, was it relevant to their life, did they learn from the session).
  Item 6 of 10: "The presenter(s) stimulated my interest in the material"
Time Frame: 48 weeks
Population: Participants providing a response to this question on the Session Evaluation Form
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 68 | 82
Participants
  Strongly agree | 50 | 54
  Agree | 14 | 26
  Disagree | 1 | 2
  Strongly Disagree | 3 | 0
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.1201, Chi-squared — [p-value comment as in outcome 21, analysis 1]

27. Secondary Outcome: Acceptability and Feasibility of Two Types of Efficacious Sexual Risk Reduction Interventions as Measured by Session Evaluation. Item 7 of 10: "The Topic of This Workshop/Session Was Relevant to my Life."
Description: Study subjects were given a brief Session Evaluation Form at the end of the behavioral intervention session consisting of ten items on a 4-point response scale aimed at eliciting information about the subject's experience with the session (i.e., was the session interesting, was it relevant to their life, did they learn from the session).
  Item 7 of 10: "The topic of this workshop/session was relevant to my life"
Time Frame: 48 weeks
Population: Participants providing a response to this question on the Session Evaluation Form
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 68 | 83
Participants
  Strongly agree | 50 | 65
  Agree | 13 | 17
  Disagree | 1 | 1
  Strongly Disagree | 4 | 0
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.1682, Chi-squared — [p-value comment as in outcome 21, analysis 1]

28. Secondary Outcome: Acceptability and Feasibility of Two Types of Efficacious Sexual Risk Reduction Interventions as Measured by Session Evaluation. Item 8 of 10: "The Workshop/Session Was Enjoyable."
Description: Study subjects were given a brief Session Evaluation Form at the end of the behavioral intervention session consisting of ten items on a 4-point response scale aimed at eliciting information about the subject's experience with the session (i.e., was the session interesting, was it relevant to their life, did they learn from the session).
  Item 8 of 10: "The workshop/session was enjoyable."
Time Frame: 48 weeks
Population: Participants providing a response to this question on the Session Evaluation Form
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 68 | 82
Participants
  Strongly agree | 47 | 49
  Agree | 14 | 28
  Disagree | 5 | 4
  Strongly Disagree | 2 | 1
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.2747, Chi-squared — [p-value comment as in outcome 21, analysis 1]

29. Secondary Outcome: Acceptability and Feasibility of Two Types of Efficacious Sexual Risk Reduction Interventions as Measured by Session Evaluation. Item 9 of 10: "I Would Recommend This Workshop/Session to Others."
Description: Study subjects were given a brief Session Evaluation Form at the end of the behavioral intervention session consisting of ten items on a 4-point response scale aimed at eliciting information about the subject's experience with the session (i.e., was the session interesting, was it relevant to their life, did they learn from the session).
  Item 9 of 10: "I would recommend this workshop/session to others."
Time Frame: 48 weeks
Population: Participants providing a response to this question on the Session Evaluation Form
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 68 | 82
Participants
  Strongly agree | 49 | 47
  Agree | 10 | 31
  Disagree | 6 | 4
  Strongly Disagree | 3 | 0
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.0046, Chi-squared — [p-value comment as in outcome 21, analysis 1]

30. Secondary Outcome: Acceptability and Feasibility of Two Types of Efficacious Sexual Risk Reduction Interventions as Measured by Session Evaluation. Item 10 of 10: "I Felt Comfortable Participating in This Workshop/Session."
Description: Study subjects were given a brief Session Evaluation Form at the end of the behavioral intervention session consisting of ten items on a 4-point response scale aimed at eliciting information about the subject's experience with the session (i.e., was the session interesting, was it relevant to their life, did they learn from the session).
  Item 10 of 10: "I felt comfortable participating in this workshop/session."
Time Frame: 48 weeks
Population: Participants providing a response to this question on the Session Evaluation Form
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 68 | 83
Participants
  Strongly agree | 54 | 55
  Agree | 9 | 23
  Disagree | 2 | 5
  Strongly Disagree | 3 | 0
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.0290, Chi-squared — [p-value comment as in outcome 21, analysis 1]

31. Secondary Outcome: Demographic and/or Behavioral Difference Between Study Groups. Behavioral Disinhibition/Risk Compensation Endpoints Will be Compared. (Age)
Description: Explores potential demographic and/or behavioral differences between youth who stay on PrEP compared to those who discontinue use.
  PrEP status (On/Off PrEP) is determined by whether a subject prematurely discontinued from the study agent or not.
  This item concerns the subject's age at enrollment.
Time Frame: 48 weeks
Population: Enrolled subjects
Measure: Mean (Standard Deviation); unit: years
Groups:
- On Prep: Remained on study agent
- Off Prep: Prematurely discontinued from the study agent
Arm/Group | On Prep | Off Prep
Number analyzed (Participants) | 141 | 59
years | 20.28 (1.32) | 19.93 (1.36)
Statistical Analysis 1: Comparison: On Prep vs Off Prep; Test type: Other; p = 0.1070, Kruskal-Wallis

32. Secondary Outcome: Explore Potential Demographic and/or Behavioral Differences Between Youth Who Are Interested in Participating in a PrEP Study Versus Those Who Are Not. Behavioral Disinhibition/Risk Compensation Endpoints Will be Compared.
Time Frame: 48 weeks
Population: Data not collected
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

33. Secondary Outcome: Demographic and/or Behavioral Difference Between Study Groups. Behavioral Disinhibition/Risk Compensation Endpoints Will be Compared. (Race, 5 Categories)
Description: Explores potential demographic and/or behavioral differences between youth who stay on PrEP compared to those who discontinue use.
  PrEP status (On/Off PrEP) is determined by whether a subject prematurely discontinued from the study agent or not.
  This item concerns the subject's race (5 categories)
Time Frame: 48 weeks
Population: Enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | On Prep | Off Prep
Number analyzed (Participants) | 141 | 59
Participants
  Asian/Pacific Islander | 2 | 0
  Black/African American | 71 | 22
  White | 25 | 17
  White/Hispanic | 15 | 6
  Other/Mixed Race | 28 | 14
Statistical Analysis 1: Comparison: On Prep vs Off Prep; Test type: Other; p = 0.2991, Fisher Exact — The chi-squared test of homogeneity is used to assess whether the proportions of the independent variable (participant self-identified race) differ between groups (On PrEP vs. Off PrEP)

34. Secondary Outcome: Demographic and/or Behavioral Difference Between Study Groups. Behavioral Disinhibition/Risk Compensation Endpoints Will be Compared. (Race, 2 Categories)
Description: Explores potential demographic and/or behavioral differences between youth who stay on PrEP compared to those who discontinue use.
  PrEP status (On/Off PrEP) is determined by whether a subject prematurely discontinued from the study agent or not.
  This item concerns the subject's race (2 categories)
Time Frame: 48 weeks
Population: Enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | On Prep | Off Prep
Number analyzed (Participants) | 141 | 59
Participants
  Black/African-American | 84 | 25
  Non-Black/African-American | 57 | 34
Statistical Analysis 1: Comparison: On Prep vs Off Prep; Test type: Other; p = 0.0298, Fisher Exact — [p-value comment as in outcome 33, analysis 1]

35. Secondary Outcome: Demographic and/or Behavioral Difference Between Study Groups. Behavioral Disinhibition/Risk Compensation Endpoints Will be Compared. (Ethnicity, Hispanic vs. Non-Hispanic or Latino)
Description: Explores potential demographic and/or behavioral differences between youth who stay on PrEP compared to those who discontinue use.
  PrEP status (On/Off PrEP) is determined by whether a subject prematurely discontinued from the study agent or not.
  This item concerns the subject's ethnicity, (Hispanic vs. Non-Hispanic or Latino)
Time Frame: 48 weeks
Population: Enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | On Prep | Off Prep
Number analyzed (Participants) | 141 | 59
Participants
  Hispanic or Latino | 36 | 17
  Non-Hispanic | 103 | 42
  Refused to answer | 2 | 0
Statistical Analysis 1: Comparison: On Prep vs Off Prep; Test type: Other; p = 0.8643, Fisher Exact — The chi-squared test of homogeneity is used to assess whether the proportions of the independent variable (participant self-identified ethnicity) differ between groups (On PrEP vs. Off PrEP)

36. Secondary Outcome: Demographic and/or Behavioral Difference Between Study Groups. Behavioral Disinhibition/Risk Compensation Endpoints Will be Compared. (BMI, Categorical)
Description: Explores potential demographic and/or behavioral differences between youth who stay on PrEP compared to those who discontinue use.
  PrEP status (On/Off PrEP) is determined by whether a subject prematurely discontinued from the study agent or not.
  This item concerns the subject's BMI (kg/m2), assessed categorically.
Time Frame: 48 weeks
Population: Enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | On Prep | Off Prep
Number analyzed (Participants) | 141 | 59
Participants
  Underweight (<18.5) | 6 | 3
  Normal (18.5- <25) | 78 | 31
  Overweight (25.0 - <30) | 31 | 12
  Obese (>=30) | 26 | 13
Statistical Analysis 1: Comparison: On Prep vs Off Prep; Test type: Other; p = 0.9037, Fisher Exact — The chi-squared test of homogeneity is used to assess whether the proportions of the independent variable (participant BMI) differ between groups (On PrEP vs. Off PrEP)

37. Secondary Outcome: Demographic and/or Behavioral Difference Between Study Groups. Behavioral Disinhibition/Risk Compensation Endpoints Will be Compared. (Log 10 Viral Load)
Description: Explores potential demographic and/or behavioral differences between youth who stay on PrEP compared to those who discontinue use.
  PrEP status (On/Off PrEP) is determined by whether a subject prematurely discontinued from the study agent or not.
  This item concerns the subject's viral load, assessed here as Log 10 Viral Load (copies/ml)
Time Frame: 48 weeks
Population: Enrolled subjects
Measure: Mean (Standard Deviation); unit: copies/ml
Arm/Group | On Prep | Off Prep
Number analyzed (Participants) | 141 | 59
copies/ml | 1.22 (0.60) | 1.14 (0.15)
Statistical Analysis 1: Comparison: On Prep vs Off Prep; Test type: Other; p = 0.5279, Kruskal-Wallis

38. Secondary Outcome: Demographic and/or Behavioral Difference Between Study Groups. Behavioral Disinhibition/Risk Compensation Endpoints Will be Compared. (High Risk Sex Acts)
Description: Explores potential demographic and/or behavioral differences between youth who stay on PrEP compared to those who discontinue use.
  PrEP status (On/Off PrEP) is determined by whether a subject prematurely discontinued from the study agent or not.
  This item concerns whether the subject reported any high risk sex acts with a male partner, defined as an answer of greater than 0 to the question "Of these males (male partners), how many did you have unprotected oral or anal sex with since the last time you took this survey?"
Time Frame: 48 weeks
Population: Participants providing ACASI data for these questions
Measure: Count of Participants; unit: Participants
Arm/Group | On Prep | Off Prep
Number analyzed (Participants) | 123 | 54
Participants
  Yes (Had high risk sex acts w/ male partner) | 101 | 42
  No (no high risk sex acts w/ male partner) | 22 | 12
Statistical Analysis 1: Comparison: On Prep vs Off Prep; Test type: Other; p = 0.5369, Fisher Exact — The chi-squared test of homogeneity is used to assess whether the proportions of the independent variable (participation in high-risk sex acts) differ between groups (On PrEP vs. Off PrEP)

39. Secondary Outcome: Acceptability and Feasibility of Text Message Reminders: Number Using Text Messaging Reminders
Description: Total number of subjects who signed up for text message reminders
Time Frame: 48 weeks
Population: This objective did not involve comparison of the behavioral intervention groups. All participants in both groups received FTC/TDF (Truvada®) and were eligible to receive text messages. As a result, this outcome was not assessed separately for each group.
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 200
Participants | 76

40. Secondary Outcome: Acceptability and Feasibility of Text Message Reminders: Number Discontinuing Text Messaging Reminders
Description: Number of subjects who discontinued receiving text message reminders while they were still on the study agent
Time Frame: 48 weeks
Population: Total number of subjects signed up for text message reminders This objective did not involve comparison of the behavioral intervention groups. All participants in both groups received FTC/TDF (Truvada®) and were eligible to receive text messages. As a result, this outcome was not assessed separately for each group.
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 76
Participants | 3

41. Secondary Outcome: Acceptability and Feasibility of Text Message Reminders as Measured by Subject Rating of the Reasons for Missing Medications on a 4-point Likert Scale. (Question 1: Away From Home)
Description: Subjects were asked to rate various measures as "Never," "Rarely," "Sometimes," or "Often" the reason for missing taking study pills. Data shown for Week 48.
  Question: In the past month, how often have you missed taking your study pills because you:
  "Were away from home?"
Time Frame: 48 weeks
Population: Participants enrolled at Week 48 providing a response to this question.
Measure: Count of Participants; unit: Participants
Groups:
- PCC Behavioral Intervention Group: PCC Behavioral Intervention combined with open label FTC/TDF (Truvada®) as PrEP
  PCC: Personalized Cognitive Counseling (PCC) is based on the Model of Relapse Prevention and Gold's Self-Appraisal of Risk Behavior. PCC is a 1-hour, single-session, individual level intervention administered by a trained counselor in a clinic setting.
  Emtricitabine/tenofovir (FTC/TDF (Truvada®)): All subjects will be provided with daily FTC/TDF (Truvada®) as Pre-exposure prophylaxis
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 74 | 49
Participants
  Never | 31 | 22
  Rarely | 17 | 11
  Sometimes | 19 | 10
  Often | 7 | 6
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.2193, Chi-squared — The chi-squared test of homogeneity is used to assess whether the proportions of the independent variable (participant responses to this question) differ between intervention arms

42. Secondary Outcome: Acceptability and Feasibility of Text Message Reminders as Measured by Subject Rating of the Reasons for Missing Medications on a 4-point Likert Scale. (Question 2: Busy With Other Things)
Description: Subjects were asked to rate various measures as "Never," "Rarely," "Sometimes," or "Often" the reason for missing taking study pills. Data shown for Week 48.
  Question: In the past month, how often have you missed taking your study pills because you:
  "Were too busy with other things?"
Time Frame: 48 weeks
Population: Participants enrolled at Week 48 providing a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 74 | 49
Participants
  Never | 33 | 24
  Rarely | 17 | 10
  Sometimes | 14 | 11
  Often | 10 | 4
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.1255, Chi-squared — [p-value comment as in outcome 41, analysis 1]

43. Secondary Outcome: Acceptability and Feasibility of Text Message Reminders as Measured by Subject Rating of the Reasons for Missing Medications on a 4-point Likert Scale. (Question 3: Simply Forgot)
Description: Subjects were asked to rate various measures as "Never," "Rarely," "Sometimes," or "Often" the reason for missing taking study pills. Data shown for Week 48.
  Question: In the past month, how often have you missed taking your study pills because you:
  "Simply forgot?"
Time Frame: 48 weeks
Population: Participants enrolled at Week 48 providing a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 74 | 49
Participants
  Never | 28 | 21
  Rarely | 18 | 14
  Sometimes | 18 | 9
  Often | 10 | 5
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.0706, Chi-squared — [p-value comment as in outcome 41, analysis 1]

44. Secondary Outcome: Acceptability and Feasibility of Text Message Reminders as Measured by Subject Rating of the Reasons for Missing Medications on a 4-point Likert Scale. (Question 4: Too Many Pills)
Description: Subjects were asked to rate various measures as "Never," "Rarely," "Sometimes," or "Often" the reason for missing taking study pills. Data shown for Week 48.
  Question: In the past month, how often have you missed taking your study pills because you:
  "Had too many study pills to take?"
Time Frame: 48 weeks
Population: Participants enrolled at Week 48 providing a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 73 | 49
Participants
  Never | 62 | 46
  Rarely | 7 | 1
  Sometimes | 2 | 1
  Often | 2 | 1
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.0088, Chi-squared — [p-value comment as in outcome 41, analysis 1]

45. Secondary Outcome: Acceptability and Feasibility of Text Message Reminders as Measured by Subject Rating of the Reasons for Missing Medications on a 4-point Likert Scale. (Question 5: Side Effects)
Description: Subjects were asked to rate various measures as "Never," "Rarely," "Sometimes," or "Often" the reason for missing taking study pills. Data shown for Week 48.
  Question: In the past month, how often have you missed taking your study pills because you:
  "Wanted to avoid side effects?"
Time Frame: 48 weeks
Population: Participants enrolled at Week 48 providing a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 73 | 49
Participants
  Never | 64 | 42
  Rarely | 7 | 4
  Sometimes | 2 | 1
  Often | 0 | 2
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.2482, Chi-squared — [p-value comment as in outcome 41, analysis 1]

46. Secondary Outcome: Acceptability and Feasibility of Text Message Reminders as Measured by Subject Rating of the Reasons for Missing Medications on a 4-point Likert Scale. (Question 6: Others Notice)
Description: Subjects were asked to rate various measures as "Never," "Rarely," "Sometimes," or "Often" the reason for missing taking study pills. Data shown for Week 48.
  Question: In the past month, how often have you missed taking your study pills because you:
  "Did not want others to notice you taking meds?"
Time Frame: 48 weeks
Population: Participants enrolled at Week 48 providing a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 74 | 49
Participants
  Never | 65 | 43
  Rarely | 7 | 3
  Sometimes | 1 | 1
  Often | 1 | 2
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.1647, Chi-squared — [p-value comment as in outcome 41, analysis 1]

47. Secondary Outcome: Acceptability and Feasibility of Text Message Reminders as Measured by Subject Rating of the Reasons for Missing Medications on a 4-point Likert Scale. (Question 7: Routine Change)
Description: Subjects were asked to rate various measures as "Never," "Rarely," "Sometimes," or "Often" the reason for missing taking study pills. Data shown for Week 48.
  Question: In the past month, how often have you missed taking your study pills because you:
  "Had a change in daily routine?"
Time Frame: 48 weeks
Population: Participants enrolled at Week 48 providing a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 74 | 49
Participants
  Never | 51 | 31
  Rarely | 9 | 5
  Sometimes | 10 | 7
  Often | 4 | 6
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.6880, Chi-squared — [p-value comment as in outcome 41, analysis 1]

48. Secondary Outcome: Acceptability and Feasibility of Text Message Reminders as Measured by Subject Rating of the Reasons for Missing Medications on a 4-point Likert Scale. (Question 8: Study Pill Harmful)
Description: Subjects were asked to rate various measures as "Never," "Rarely," "Sometimes," or "Often" the reason for missing taking study pills. Data shown for Week 48.
  Question: In the past month, how often have you missed taking your study pills because you:
  "Felt like the study pill was toxic/harmful?"
Time Frame: 48 weeks
Population: Participants enrolled at Week 48 providing a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 74 | 49
Participants
  Never | 71 | 45
  Rarely | 3 | 1
  Sometimes | 0 | 1
  Often | 0 | 2
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.2881, Chi-squared — [p-value comment as in outcome 41, analysis 1]

49. Secondary Outcome: Acceptability and Feasibility of Text Message Reminders as Measured by Subject Rating of the Reasons for Missing Medications on a 4-point Likert Scale. (Question 9: Fell Asleep)
Description: Subjects were asked to rate various measures as "Never," "Rarely," "Sometimes," or "Often" the reason for missing taking study pills. Data shown for Week 48.
  Question: In the past month, how often have you missed taking your study pills because you:
  "Fell asleep/slept through dose time?"
Time Frame: 48 weeks
Population: Participants enrolled at Week 48 providing a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 74 | 49
Participants
  Never | 52 | 35
  Rarely | 13 | 6
  Sometimes | 5 | 7
  Often | 4 | 1
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.2223, Chi-squared — [p-value comment as in outcome 41, analysis 1]

50. Secondary Outcome: Acceptability and Feasibility of Text Message Reminders as Measured by Subject Rating of the Reasons for Missing Medications on a 4-point Likert Scale. (Question 10: Felt Ill)
Description: Subjects were asked to rate various measures as "Never," "Rarely," "Sometimes," or "Often" the reason for missing taking study pills. Data shown for Week 48.
  Question: In the past month, how often have you missed taking your study pills because you:
  "Felt sick or ill?"
Time Frame: 48 weeks
Population: Participants enrolled at Week 48 providing a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 74 | 49
Participants
  Never | 61 | 43
  Rarely | 9 | 1
  Sometimes | 3 | 4
  Often | 1 | 1
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.0617, Chi-squared — [p-value comment as in outcome 41, analysis 1]

51. Secondary Outcome: Acceptability and Feasibility of Text Message Reminders as Measured by Subject Rating of the Reasons for Missing Medications on a 4-point Likert Scale. (Question 11: Felt Depressed)
Description: Subjects were asked to rate various measures as "Never," "Rarely," "Sometimes," or "Often" the reason for missing taking study pills. Data shown for Week 48.
  Question: In the past month, how often have you missed taking your study pills because you:
  "Felt depressed/overwhelmed?"
Time Frame: 48 weeks
Population: Participants enrolled at Week 48 providing a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 74 | 49
Participants
  Never | 62 | 43
  Rarely | 10 | 1
  Sometimes | 1 | 4
  Often | 1 | 1
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.0868, Chi-squared — [p-value comment as in outcome 41, analysis 1]

52. Secondary Outcome: Acceptability and Feasibility of Text Message Reminders as Measured by Subject Rating of the Reasons for Missing Medications on a 4-point Likert Scale. (Question 12: Ran Out of Pills)
Description: Subjects were asked to rate various measures as "Never," "Rarely," "Sometimes," or "Often" the reason for missing taking study pills. Data shown for Week 48.
  Question: In the past month, how often have you missed taking your study pills because you:
  "Ran out of study pills?"
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 74 | 49
Participants
  Never | 67 | 44
  Rarely | 7 | 1
  Sometimes | 0 | 1
  Often | 0 | 3
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.1847, Chi-squared — [p-value comment as in outcome 41, analysis 1]

53. Secondary Outcome: Acceptability and Feasibility of Text Message Reminders as Measured by Subject Rating of the Reasons for Missing Medications on a 4-point Likert Scale. (Question 13: No Risky Sex)
Description: Subjects were asked to rate various measures as "Never," "Rarely," "Sometimes," or "Often" the reason for missing taking study pills. Data shown for Week 48.
  Question: In the past month, how often have you missed taking your study pills because you:
  "Didn't think you needed it because you weren't having risk sex?"
Time Frame: 48 weeks
Population: Participants enrolled at Week 48 providing a response to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
Number analyzed (Participants) | 73 | 49
Participants
  Never | 58 | 43
  Rarely | 12 | 4
  Sometimes | 1 | 1
  Often | 2 | 1
Statistical Analysis 1: Comparison: 3MV Behavioral Intervention Group vs PCC Behavioral Intervention Group; Test type: Other; p = 0.0226, Chi-squared — [p-value comment as in outcome 41, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the duration of the project, from the start of enrollment on 11/21/2012 until study follow-up completion on 11/7/2015. All enrolled participants were assessed over the course of visits through Week 48, and a subset of participants meeting eligibility requirements were followed for an additional 48 weeks.
Description: Per protocol, only grade 3 and higher clinical adverse events and lab toxicities are systematically recorded on the Adverse Event Evaluation form and reported here.
Arm/Group | 3MV Behavioral Intervention Group | PCC Behavioral Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/72
Serious Adverse Events (participants affected / at risk) | 7/128 | 1/72
Other Adverse Events (participants affected / at risk) | 10/128 | 4/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3MV Behavioral Intervention Group (N=128) | PCC Behavioral Intervention Group (N=72)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 2 (3) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3MV Behavioral Intervention Group (N=128) | PCC Behavioral Intervention Group (N=72)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 1 (1)
Cytomegalovirus Hepatitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Shigella (Infections and infestations) | 1 (1) | 0 (0)
Avulsion Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Decreased appetitie (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Testicular Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Adolescent Medicine Trials Network (ATN) for HIV/AIDS Interventions Publication Policy outlines procedures for the development and review of abstracts, publications, and presentations. The Adolescent Medicine Leadership Group (AMLG) retains custody of and primary rights to the data. Use of data must be approved by the protocol team and AMLG.